CLINICAL TRIAL: NCT00472706
Title: A Randomized Clinical Trial of Excision Versus Photodynamic Therapy in Bowen's Disease
Brief Title: Trial of Excision Versus Photodynamic Therapy in the Treatment of Bowen's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped because of disappointing inclusion rates
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Drs. A. Verzijl, Catharina hospital/Erasmus MC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06-16107
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Bowen's Disease
Keywords: Treatment; Excision; Photodynamic therapy; Recurrence rate; Cosmetic outcome
MeSH Terms: conditions — Bowen's Disease | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Excision
  Interventions: Procedure: excision
- 2 (Active Comparator): Photodynamic therapy
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: excision — excision 3 mm margin
  Arms: 1
Procedure: Photodynamic therapy — Photodynamic therapy
  Arms: 2

SUMMARY:
The purpose of this study is to identify the most optimal therapy for Bowen's disease: excision versus Photodynamic therapy.

DETAILED DESCRIPTION:
The study is a randomized clinical trial in which two treatment options for Bowen's disease, excision and photodynamic therapy, are compared on recurrence rate, cosmesis en expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histological proven Bowen's disease on scalp, face, trunk, arms and legs
* Informed Consent

Exclusion Criteria:

* Recurrent Bowen's disease
* Anogenital or subungual Bowe's disease
* Other skin malignancy in the same area
* Porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Estimated); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
recurrence rate | two years

SECONDARY OUTCOMES:
cosmetic outcome | one year

CONTACTS AND LOCATIONS:
Overall Officials: Annette Verzijl, MD, Principal Investigator — Catharina hospital/Erasmus MC